CLINICAL TRIAL: NCT03459079
Title: Efficacy, Safety and Mechanism of Action of Lanifibranor (IVA337) in Patients With Type 2 Diabetes and Nonalcoholic Fatty Liver Disease
Brief Title: Lanifibranor in Patients With Type 2 Diabetes & Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Inventiva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201800838 -A; PRO00018845 AGR00010853 (Other: University of Florida); OCR17599 (Other: Universiy of Florida)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD); Type 2 Diabetes (T2DM)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — lanifibranor

STUDY DESIGN:
Intervention Model Description: A two arm randomized (1:1), double-blind, placebo-controlled, trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- lanifibranor arm (Active Comparator): Two arm, randomized (1:1), double-blind, placebo-controlled, 24-week treatment study receiving lanifibranor 800 mg/day.
  Interventions: Drug: Lanifibranor
- Placebo (Placebo Comparator): Two arm, randomized (1:1), double-blind, placebo-controlled, 24-week treatment study receiving placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lanifibranor — The film-coated tablet contains 400 mg of the active ingredient lanifibranor (IVA337) for an immediate release formulation. Participants receive 800mg/ day
  Other Names: IVA 337
  Arms: lanifibranor arm
Other: Placebo — Film-coated tablets with a core containing 900 mg of a physical mixture of lactose monohydrate, microcrystalline cellulose, pre-gelatinized starch and magnesium stearate serve as placebo.
  Arms: Placebo

SUMMARY:
The primary aim is to establish the safety, efficacy and mechanism of action of lanifibranor in patients with type 2 diabetes (T2DM) and nonalcoholic fatty liver disease (NAFLD). Specifically, to determine if lanifibranor decreases intrahepatic triglycerides (IHTG) (primary endpoint), improves hepatic insulin sensitivity, endogenous (hepatic) glucose production, de novo lipogenesis (DNL), HbA1c and lipid profiles. In addition, exploratory analysis with surrogate plasma biomarkers and imaging on liver fibrosis changes on with treatment will be performed.

DETAILED DESCRIPTION:
The study is a two-arm (placebo, lanifibranor 800 mg/day), randomized (1:1), double-blind, placebo-controlled, 24-week treatment study. Thirty four (n=34)patients with T2DM will be randomized, allowing for a 10% drop-out rate. The diagnosis of NAFLD on imaging will be done by measuring IHTG using the gold-standard magnetic resonance and spectroscopy (¹H-MRS) technique. Ten non-diabetic subjects without NAFLD will also serve as a control group for the metabolic and imaging procedures. The study will last 34-36 weeks (~6-8 weeks for run-in, 24 weeks of treatment and 4 weeks post-study follow-up), with an estimated recruitment period of ~9 months. Patients with uncontrolled T2DM and a diagnosis of "fatty liver" per history (elevated AST/ALT and/or liver fat on liver ultrasound or ¹H-MRS and/or other appropriate imaging technique - see below). Participants may be treated by diet only, or be on a stable dose of metformin and/or a sulfonylurea and/or a DPP-IV inhibitor for ≥ 2 months prior to enrollment. If the HbA1c is ≤8.0% on any of these diabetes medications, the dose of these medications will be kept stable throughout the study and baseline studies performed as outlined below. If the HbA1c is > 8.0% but ≤ 9.5%, metformin (minimum dose required: 1,000 mg/day for metformin) and/or a sulfonylurea (minimum dose required: glimepiride 2 mg once daily) will be added, or doses maximized, during the first 2 weeks of the lead-in period. Afterwards, patient's metformin or sulfonylurea dose will be maintained at the new dose stable for 4 weeks before baseline metabolic and study-specific liver imaging.

After patients sign the informed consent and meet eligibility criteria, baseline imaging and metabolic studies will be performed. These will include measurement of IHTG by 1H-MRS, liver fibrosis by VCTE (Fibroscan) and MRE, and additional imaging by T1 MRI mapping. Metabolic testing will be done with the patient being admitted to the CRC (clinical research unit) for an overnight stay. Assessment of insulin sensitivity and DNL will be done with the administration of stable isotopes of glucose (intravenously) and deuterium labeled water (orally) to measure glucose and lipid turnover and substrate oxidation (with indirect calorimetry) during a euglycemic hyperinsulinemic clamp.

After all baseline tests are completed, patients will be asked to take a therapeutic dose of 800 mg lanifibranor (QD), or placebo, for 24 weeks. They will be closely followed by study staff every 4 weeks with visits to the CRC and interim phone calls. At 24 weeks, all baseline tests will be repeated and treatment considered completed. There will be a final, off-drug, safety follow-up visit 4 weeks after treatment at week 28. After this the participant will have completed all study procedures.

Note: The investigators recalculated the sample size for the primary endpoint of change in intrahepatic triglyceride (IHTG) measured by 1H-MRS with lanifibranor (800 mg/day) vs. placebo based on the data from the population with diabetes from the Phase IIb NATIVE (NCT03008070: NAsh Trial to Validate IVA337 Efficacy; liver histology results) and comparing to prior studies by Dr. Cusi et al that had simultaneous liver histology and liver fat measured by 1H-MRS (Belfort et al, NEJM 2006; Cusi et al, Annals Int Med 2016). From this analysis, the required sample size per group calls for 15 patients in each arm (lanifibranor vs. placebo) to complete treatment. Conservatively assuming that 10 % of the randomized patients will not complete the trial (dropouts), the total number of patients to be randomized is 33-34 patients.

ELIGIBILITY:
Inclusion Criteria:

* Be able to communicate meaningfully with the investigator and legally competent to provide written informed consent
* Have an age between 21 to 75 years inclusive
* Subjects should be on stable standard of care and background therapy for ongoing chronic conditions, including stable doses of anti-diabetic medications, for at least two (2) months prior to trial entry
* Have uncontrolled diabetes with a fasting plasma glucose (FPG) ≥ 100 mg/dL but ≤ 250 mg/dL and HbA1c ≥ 6.0% but ≤ 9.5%, on diet alone, or on metformin (≥1,000 mg/day), and/or sulfonylurea and/or DPP-IV therapy, SGLT2 inhibitors or GLP1RA. These medicines will be continued at stable doses during the entire study.

  1. Subjects with an HbA1c > 8.0% but ≤ 9.5% will have their metformin (minimum dose required: 1,000 mg/day) maximized to 1,000 mg BID and/or glimepiride 2 mg once daily added during the first 2 weeks of the run-in period. The baseline visit to initiate lanifibranor (V4; Time 0 or randomization visit) will be not sooner than 8 weeks from diabetes medication titration and the patient should have an HbA1c ≤9.0% to proceed to randomization (V4).
  2. In addition, if both metformin and glimepiride (or another sulfonylurea) are already maximized at study entry (or the patient is intolerant to either) and the HbA1c ≥ 9.0% but ≤9.5%, we will add sitagliptin 100 mg daily (or an equivalent dose of another DPP-IV inhibitor) to reach an HbA1c ≤9.0% to proceed to randomization (V4).
* Presence of hepatic steatosis (Intrahepatic Triglycerides IHTG) > 10 % determined by Magnetic Resonance and Spectroscopy (1H-MRS).
* Have no new symptoms associated with decompensated diabetes in the previous 3 months.
* Compensated liver disease with the following hematologic and biochemical criteria on entry into protocol:

  * Hemoglobin > 11 g/dL for females and > 12 g/dL for males
  * White blood cell (WBC) > 2.5 K/µL
  * Neutrophil count > 1.5 K/µL
  * Total bilirubin ≤ 1.3 mg/dL (≤ 22.2 µmol/L). Patients with bilirubin ≤ 1.3 mg/dL can be included if non-conjugated bilirubin in the setting of a Gilbert's syndrome.
  * Albumin > 36 g/L
* No other causes of chronic liver disease (autoimmune, primary biliary cholangitis, HBV, HCV, Wilson's, α-1-antitrypsin deficiency, hemochromatosis, other).
* Negative pregnancy test or at least two-year post-menopausal. Women with childbearing potential (i.e. fertile, following menarche and until becoming post- menopausal unless permanently sterile) must be using a highly effective method of contraception (i.e. combined (estrogen and progesterone containing) hormonal/ progesterone-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner). The contraceptive method will have to be followed for at least one menstruation cycle after the end of the study.

Exclusion Criteria:

* Evidence of liver disease other than NAFLD.
* History of excessive alcohol intake, defined by ≥ 21 units of alcohol per week in males and ≥14 units of alcohol per week in females for two years prior to enrollment, where a "unit" of alcohol is equivalent to 12-ounce beer, 4-ounce glass of wine, or 1 ounce shot of hard liquor.
* Unstable metabolic condition: Weight change > 5 kg in the 3 months prior to enrollment, diabetes with poor glycemic control (HgbA1c > 9.5% or FPG > 250 mg/dl), introduction of an anti-obesity drug/malabsorptive or restrictive bariatric (weight loss) surgery in the past 6 months prior to screening.
* History of gastrointestinal malabsorptive bariatric surgery within less than 5 years or ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.
* Subjects on sulfonylureas, metformin, GLP-1RA or DPP-IV unless the dose and body weight (within 5%) have been stable for at least two (2) months prior to study entry.
* Patients on insulin, pioglitazone (or prior use in the past 12 months).
* Patients on any of the following medications unless the patient has been on stable doses of such agents for the past two (2) months before entry into the study: thiazide or furosemide diuretics, beta- blockers, or other chronic medications with known adverse effects on glucose tolerance levels. Patients may be taking stable doses of estrogens or other hormonal replacement therapy if the patient has been on these agents for the prior two (2) months. Patients taking systemic glucocorticoids will be excluded.

Treatment with strong inducers or inhibitors of CYP2C8, or treatment with substrates of CYP2B6 or CYP2C8. When administered chronically, they should be replaced 2 months before trial entry (See Inclusion criterion #3). If not administered chronically, they should be stopped at least 7 days before first dosing.

-Patients with:

1. History of myopathies or evidence of active muscle diseases
2. Unstable cardiovascular disease, including:

i. Unstable angina (i.e., new or worsening symptoms of coronary heart disease within the past 3 months), acute coronary syndrome within the past 6 months, acute myocardial infarction in the past 3 months or heart failure of New York Heart Association class (III-IV) or worsening congestive heart failure, or coronary artery intervention, within the past 6 months ii. History of (within prior 3 months) or current unstable cardiac dysrhythmias iii. Uncontrolled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg.

iv. Stroke or transient ischemic attack within the prior 6 months c. History of malignancy in the past 5 years and/or active neoplasm with the exception of resolved superficial nonmelanoma skin cancer d. History of bladder disease and/or hematuria or has current hematuria unless due to a urinary tract infection e. Any of the following laboratory values: ii. Serum bilirubin > 1.3 mg/dL (or > 22.2 µmol/L). Patients with bilirubin >1.3 mg/dL can be included if non-conjugated bilirubin in the setting of a Gilbert's syndrome.

iii. Serum ALT > 3X ULN iv. INR > 1.2 v. Platelets < 150,000 per microliter of blood vi. Renal impairment as demonstrated by estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2 vii. Total creatinine kinase > 1.5 X ULN viii. Lipase > 1.3X ULN or >2.0X ULN if on a DPP-IV inhibitor. *(if abnormal values are confirmed when repeated within 3 weeks) ix. Hemoglobin A1c > 9.5%

* Significant systemic or major illnesses other than liver disease, including those listed in exclusion criteria #8 and pulmonary disease, organ transplantation, serious psychiatric disease, that, in the opinion of the investigator, would preclude treatment with lanifibranor and/or adequate follow up.
* HB antigen > 0, HCV > 0 (patients with a history of HCV infection can be included if HCV PCR is negative since more than 3 years), prior history of HIV infection.
* Pregnancy/lactation or inability to adhere to adequate contraception in women of child-bearing potential.
* Any other condition which, in the opinion of the investigator would impede competence or compliance or possibly hinder completion of the study.
* Body mass index (BMI) > 45 kg/m2.
* Type 1 diabetes and type 2 diabetic patient on insulin.
* Diabetic ketoacidosis.
* Fasting plasma triglycerides > 500 mg/dL.
* Hemostasis disorders or current treatment with anticoagulants.
* Participation in any other investigational drug study within the previous 3 months.
* Have a known hypersensitivity to any of the ingredients or excipients of the IMP including: Lactose monohydrate, hypromellose, sodium lauryl sulphate, sodium starch glycolate, magnesium stearate, Opadry™ II 85F18422, DSS Granular, cellulose microcrystalline, maize starch.
* Be possibly dependent on the Investigator (e.g., including, but not limited to, affiliated employee).
* Osteopenia or any other well documented bone disease. Patient without well documented osteopenia treated with vitamin D and/or calcium based supplements for preventive reasons can be included.
* Claustrophobia to a degree that prevents tolerance of MRI scanning procedure. Sedation is permitted at discretion of investigator.
* Metallic implant of any sort that prevents MRI examination including, but not limited to: aneurysm clips, metallic foreign body, vascular grafts or cardiac implants, neural stimulator, metallic contraceptive device, tattoo, body piercing that cannot be removed, cochlear implant; or any other contraindication to MRI examination.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cusi, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Belfort R, Harrison SA, Brown K, Darland C, Finch J, Hardies J, Balas B, Gastaldelli A, Tio F, Pulcini J, Berria R, Ma JZ, Dwivedi S, Havranek R, Fincke C, DeFronzo R, Bannayan GA, Schenker S, Cusi K. A placebo-controlled trial of pioglitazone in subjects with nonalcoholic steatohepatitis. N Engl J Med. 2006 Nov 30;355(22):2297-307. doi: 10.1056/NEJMoa060326. PMID 17135584
- [Background] Cusi K, Orsak B, Bril F, Lomonaco R, Hecht J, Ortiz-Lopez C, Tio F, Hardies J, Darland C, Musi N, Webb A, Portillo-Sanchez P. Long-Term Pioglitazone Treatment for Patients With Nonalcoholic Steatohepatitis and Prediabetes or Type 2 Diabetes Mellitus: A Randomized Trial. Ann Intern Med. 2016 Sep 6;165(5):305-15. doi: 10.7326/M15-1774. Epub 2016 Jun 21. PMID 27322798
- [Background] Cusi K. Role of obesity and lipotoxicity in the development of nonalcoholic steatohepatitis: pathophysiology and clinical implications. Gastroenterology. 2012 Apr;142(4):711-725.e6. doi: 10.1053/j.gastro.2012.02.003. Epub 2012 Feb 8. PMID 22326434
- [Background] Lomonaco R, Bril F, Portillo-Sanchez P, Ortiz-Lopez C, Orsak B, Biernacki D, Lo M, Suman A, Weber MH, Cusi K. Metabolic Impact of Nonalcoholic Steatohepatitis in Obese Patients With Type 2 Diabetes. Diabetes Care. 2016 Apr;39(4):632-8. doi: 10.2337/dc15-1876. Epub 2016 Feb 9. PMID 26861926
- [Background] Bril F, Cusi K. Management of Nonalcoholic Fatty Liver Disease in Patients With Type 2 Diabetes: A Call to Action. Diabetes Care. 2017 Mar;40(3):419-430. doi: 10.2337/dc16-1787. PMID 28223446
- [Background] Boubia B, Poupardin O, Barth M, Binet J, Peralba P, Mounier L, Jacquier E, Gauthier E, Lepais V, Chatar M, Ferry S, Thourigny A, Guillier F, Llacer J, Amaudrut J, Dodey P, Lacombe O, Masson P, Montalbetti C, Wettstein G, Luccarini JM, Legendre C, Junien JL, Broqua P. Design, Synthesis, and Evaluation of a Novel Series of Indole Sulfonamide Peroxisome Proliferator Activated Receptor (PPAR) alpha/gamma/delta Triple Activators: Discovery of Lanifibranor, a New Antifibrotic Clinical Candidate. J Med Chem. 2018 Mar 22;61(6):2246-2265. doi: 10.1021/acs.jmedchem.7b01285. Epub 2018 Feb 27. PMID 29446942
- [Background] Wettstein G, Luccarini JM, Poekes L, Faye P, Kupkowski F, Adarbes V, Defrene E, Estivalet C, Gawronski X, Jantzen I, Philippot A, Tessier J, Tuyaa-Boustugue P, Oakley F, Mann DA, Leclercq I, Francque S, Konstantinova I, Broqua P, Junien JL. The new-generation pan-peroxisome proliferator-activated receptor agonist IVA337 protects the liver from metabolic disorders and fibrosis. Hepatol Commun. 2017 Jun 19;1(6):524-537. doi: 10.1002/hep4.1057. eCollection 2017 Aug. PMID 29404476
- [Background] Avouac J, Konstantinova I, Guignabert C, Pezet S, Sadoine J, Guilbert T, Cauvet A, Tu L, Luccarini JM, Junien JL, Broqua P, Allanore Y. Pan-PPAR agonist IVA337 is effective in experimental lung fibrosis and pulmonary hypertension. Ann Rheum Dis. 2017 Nov;76(11):1931-1940. doi: 10.1136/annrheumdis-2016-210821. Epub 2017 Aug 11. PMID 28801346
- [Background] Ruzehaji N, Frantz C, Ponsoye M, Avouac J, Pezet S, Guilbert T, Luccarini JM, Broqua P, Junien JL, Allanore Y. Pan PPAR agonist IVA337 is effective in prevention and treatment of experimental skin fibrosis. Ann Rheum Dis. 2016 Dec;75(12):2175-2183. doi: 10.1136/annrheumdis-2015-208029. Epub 2016 Mar 9. PMID 26961294
- [Derived] Barb D, Kalavalapalli S, Godinez Leiva E, Bril F, Huot-Marchand P, Dzen L, Rosenberg JT, Junien JL, Broqua P, Rocha AO, Lomonaco R, Abitbol JL, Cooreman MP, Cusi K. Pan-PPAR agonist lanifibranor improves insulin resistance and hepatic steatosis in patients with T2D and MASLD. J Hepatol. 2025 Jun;82(6):979-991. doi: 10.1016/j.jhep.2024.12.045. Epub 2025 Jan 15. PMID 39824443
- See also: Website of the Division of Endocrinology, Diabetes and Metabolism at the University of Florida — http://endocrinology.medicine.ufl.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 128 total enrolled participants, 38 subjects with type 2 diabetes met inclusion criteria and were randomized to be treated. 10 healthy controls met inclusion criteria and completed imaging and other study assessments. This study was performed during the epidemic of COVID that greatly impacted recruitment and promoted dropout.
Groups:
- Healthy Control Group (Not a Treatment Arm): This group ONLY underwent baseline labs, baseline liver fat assessment and one insulin sensitivity measurement to establish the "normal" for these parameters and to which compare the 2 treatment arms (i.e., lanifibranor and placebo arms). They are NOT treatment arms and participation ended after qualifying and the above studies.
Period: Overall Study
Arm/Group | Lanifibranor Arm | Placebo | Healthy Control Group (Not a Treatment Arm)
Started | 20 | 18 | 10
Completed | 14 | 14 | 10
Not Completed | 6 | 4 | 0
Not completed — Adverse Event | 4 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanifibranor Arm | Placebo | Healthy Control Group (Not a Treatment Arm) | Total
Number analyzed (Participants) | 20 | 18 | 10 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7) | 58 (11) | 43 (18) | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 6 | 30
  Male | 9 | 5 | 4 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 18 | 15 | 9 | 42
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 10 | 48
Intrahepatic triglyceride content [Mean (Standard Deviation); unit: %] | 21 (7) | 18 (7) | 3 (1) | 19.5 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intrahepatic Triglycerides (IHTG) Quantified by Proton Magnetic Resonance and Spectroscopy (¹H-MRS)
Description: Changes from baseline (Adjusted LS means) in absolute percent for change in intrahepatic triglycerides (IHTG) quantified by proton magnetic resonance and spectroscopy (¹H-MRS)are reported in each arms.
Time Frame: 24 weeks of treatment
Population: We report absolute change from baseline in LS mean [95% CI]
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage decrease from baseline
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
percentage decrease from baseline | -8.7 [-11.3 to -6.0] | -3.0 [-5.9 to -0.2]

2. Secondary Outcome: Percentage of Patients With a Decrease From Baseline in IHTG (Quantified by ¹H-MRS) to Week 24 of ≥ 30%.
Description: Percentage of patients with a decrease from baseline in IHTG (quantified by ¹H-MRS) to week 24 of ≥ 30% in each group.
Time Frame: 24 weeks of treatment.
Population: ≥30% reduction in IHTG
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
percentage of participants | 65 [41 to 85] | 22 [6 to 48]

3. Secondary Outcome: Percentage of Patients With NAFLD Resolution, Defined as Having ≤ 5.5% IHTG (Quantified by 1H- MRS).
Description: Percentage of patients with NAFLD resolution, defined as having ≤ 5.5% IHTG (quantified by 1H- MRS) in both arms.
Time Frame: 24 weeks of treatment.
Population: Full Analyses Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
percentage of participants | 25 [9 to 49] | 0 [0 to 19]

4. Secondary Outcome: Improvement in Hepatic Insulin Sensitivity (Hepatic Insulin Resistance Index Reported as Relative Percent Change)
Description: Changes from baseline in hepatic insulin sensitivity (Hepatic Insulin Resistance Index) as a relative percent change is presented (i.e. [24 week result- baseline result]/baseline result *100).
Time Frame: 24 weeks of treatment.
Population: Full Analyses Set
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of baseline value
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
percentage of baseline value | -26 [-37 to -14] | -7 [-19 to 4]

5. Secondary Outcome: Improvement in Adipose Tissue Insulin Sensitivity.
Description: Changes from baseline in absolute value of adipose tissue insulin resistance (ADIPO-IR) index will be compared between both arms. This is calculated using the formula below:
  Adipo-IR index = fasting serum free fatty acid concentration x fasting plasma insulin level. A higher value indicated higher insulin resistance.
Time Frame: 24 weeks of treatment.
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
index | -2.7 [-4.3 to -1.2] | -0.7 [-2.4 to 0.9]

6. Secondary Outcome: Improvement in Muscle Insulin Sensitivity (Rd).
Description: Relative percent changes from baseline in insulin-stimulated muscle glucose disposal (%) will be compared between both arms (i.e. [24 week result- baseline result]/baseline result *100).
Time Frame: 24 weeks of treatment.
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change from baseline
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
percentage change from baseline | 30 [13 to 46] | 0 [-17 to 18]

7. Secondary Outcome: Absolute Change in Glycemic Control (Hemoglobin A1c).
Description: Absolute changes from baseline will be compared between both arms (i.e., percentage at 24 weeks subtracted from the percentage at baseline).
Time Frame: 24 weeks of treatment.
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: absolute percent change from baseline
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
absolute percent change from baseline | -0.7 [-1.0 to -0.5] | -0.1 [-0.3 to 0.2]

8. Secondary Outcome: Change in Plasma HDL-C (mg/dl).
Description: Changes from baseline will be compared between both arms.
Time Frame: 24 weeks of treatment.
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: absolute change in mg/dl from baseline
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
absolute change in mg/dl from baseline | 7.6 [4.4 to 10.7] | 0.9 [-2.4 to 4.3]

9. Secondary Outcome: Changes in Hepatic Fibrosis (Liver Stiffness Measurement by Vibration Controlled Transient Elastography in kPa) on Imaging.
Description: Changes from baseline in liver stiffness measurement in kPa by vibration controlled transient elastography measured in both arms.
Time Frame: 24 weeks of treatment.
Population: Full analysis set
Measure: Least Squares Mean (95% Confidence Interval); unit: absolute change in kPa from baseline
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
absolute change in kPa from baseline | -1.49 [-2.66 to -0.31] | -0.34 [-1.57 to 0.9]

10. Secondary Outcome: Change in Plasma Biomarkers of Liver Fibrosis (Plasma Cytokeratin 18 Measured in IU/L).
Description: Absolute change (Mean ± SD) changes from baseline in plasma cytokeratin 18 (IU/L) levels in both arms.
Time Frame: 24 weeks of treatment.
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: absolute change in from baseline in IU/L
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
absolute change in from baseline in IU/L | -130.71 (164.28) | -70.21 (230.39)

11. Secondary Outcome: Changes in Hepatic Fibrosis (Liver Stiffness Measurement by Magnetic Resonance Elastography in kPa) on Imaging.
Description: Changes from baseline in liver stiffness measurement by magnetic resonance elastography is measured in both arms (absolute change in kPa from baseline).
Time Frame: 24 weeks of treatment.
Population: Two subjects in the lanifibranor group missing this measurement due to technical errors
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 18 | 18
kPa | 0.23 [0.03 to 0.42] | -0.06 [-0.25 to 0.13]

12. Secondary Outcome: Hepatic Fibrosis (Liver Stiffness Measurement by Magnetic Resonance Elastography) on Imaging.
Description: Baseline liver stiffness measurement (LSM) by magnetic resonance elastography (in kPa) in both arms.
Time Frame: Baseline measurement of liver stiffness by magnetic resonance elastography is reported in each arm.
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Lanifibranor Arm | Placebo
Number analyzed (Participants) | 20 | 18
kPa | 2.8 (0.8) | 2.5 (1.1)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Lanifibranor Arm | Placebo | Healthy Control Group (Not a Treatment Arm)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/18 | 0/10
Other Adverse Events (participants affected / at risk) | 18/20 | 17/18 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanifibranor Arm (N=20) | Placebo (N=18) | Healthy Control Group (Not a Treatment Arm) (N=10)
COVID-19 pneumonia and pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lanifibranor Arm (N=20) | Placebo (N=18) | Healthy Control Group (Not a Treatment Arm) (N=10)
Diarrhoea (Gastrointestinal disorders) | 5/19 | 3 | 0
Elevated lipase level (Gastrointestinal disorders) | 5 | 3 | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dermatological (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Decrease in eGFR (Renal and urinary disorders) | 1 | 2 | 0
Transaminitis (Hepatobiliary disorders) | 1 | 1 | 0
Hypoglycemia (Endocrine disorders) | 1 | 0 | 0
Edema (Cardiac disorders) | 1 | 0 | 0
Hyperglycemia (Endocrine disorders) | 0 | 2 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Nausea and/or vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Upset stomach (Gastrointestinal disorders) | 2 | 0 | 0
Increased appetite (Gastrointestinal disorders) | 1 | 0 | 0
Orange stools (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Abnormal thyroid test (Endocrine disorders) | 1 | 0 | 0
Hyponatremia (Renal and urinary disorders) | 0 | 1 | 0
Hypokalemia (Renal and urinary disorders) | 0 | 1 | 0
Hypecalcemia (Endocrine disorders) | 0 | 1 | 0
Lightheadedness (Nervous system disorders) | 0 | 1 | 0
Abnormal urinalysis (Renal and urinary disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Fluctuating lipase levels (Hepatobiliary disorders) | 2 | 1 | 0
Arm pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vsasovagal reaction (Cardiac disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The original number of patients to be recruited was reduced during the trial based on the results of the NATIVE study (Francque et al, N Engl J Med. 2021 Oct 21;385(17):1547-1558. doi: 10.1056/NEJMoa2036205), as explained in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/79/NCT03459079/Prot_SAP_000.pdf